CLINICAL TRIAL: NCT05807022
Title: Evaluation of the Safety and Effectiveness of Percutaneous and Transbronchial Argon-helium Cryoablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-NHLHCRF-LX-01-0202-5
Record Dates: First submitted 2023-03-09; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Administration, Cutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous or transbronchial argon-helium cryoablation (Experimental)
  Interventions: Procedure: Percutaneous or transbronchial argon-helium cryoablation

INTERVENTIONS:
Procedure: Percutaneous or transbronchial argon-helium cryoablation — The participants would undergo Percutaneous or transbronchial argon-helium cryoablation.

SUMMARY:
The goal clinical trial is to evaluation of the safety and effectiveness of percutaneous and transbronchial argon-helium cryoablation in primary lung cancer and metastatic lung cancer. The main question it aims to answer are:Evaluation of the safety and effectiveness of percutaneous and transbronchial argon-helium cryoablation.

Participants will undergo percutaneous or transbronchial argon-helium cryoablation.

ELIGIBILITY:
Inclusion Criteria:

* Primary or metastatic lung cancer with definite pathological diagnosis
* Not suitable for thoracotomy due to serious or serious lung or systemic diseases
* Peripheral lung cancer involves pleura and chest wall, and cannot be completely removed after surgery
* There are indications for surgical resection, but the patient refuses to operate
* Single tumor, maximum diameter ≤ 5cm
* Or the number of tumors ≤ 3 and the maximum diameter ≤ 3cm
* ECOG-PS score ≤ 2
* The expected survival period is more than three months
* Those who have not participated in other clinical verifications within 3 months
* Subjects voluntarily signed the informed consent form

Exclusion Criteria:

* Serious cardio-cerebral disease or other mental diseases
* Severe pulmonary fibrosis, especially drug-induced pulmonary fibrosis
* Patients with previous severe pulmonary dysfunction, pulmonary ventilation disorder and multiple pulmonary bullae
* Have a history of immunodeficiency, including HIV test (enzyme-linked immunosorbent assay and Western blotting) positive
* Chemotherapy, radiotherapy, interventional therapy, ablation and surgical treatment within 30 days before surgical treatment
* There is a tendency to severe bleeding, and the platelet is less than 50 × 109/L and severe disorder of coagulation function
* Coagulation index (PT, TT, APTT)>2.5 times of the upper normal limit
* Malignant pleural effusion on the same side of the ablation focus was not well controlled
* Poor general condition, multiple organ failure, cachexia, severe anemia and nutritional metabolism disorder
* Those who have extensive extrapulmonary metastasis and are not suitable for ablation treatment
* Those who often use sedatives, sleeping pills, tranquilizers or other addictive drugs
* Pregnant or lactating women
* Those who can not judge the curative effect
* Other conditions determined by the researcher to be unsuitable for the group, such as inability to tolerate cryoablation, difficulty in follow-up, and other serious diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate and effective rate of target lesions | during the operation of argon-helium cryoablation
  Enhanced imaging examination (CT, MRI or color Doppler ultrasound)
Complete response rate and effective rate of target lesions | 1 week after the operation of argon-helium cryoablation
  Enhanced imaging examination (CT, MRI or color Doppler ultrasound)
Complete response rate and effective rate of target lesions | 4 weeks(±7d) after the operation of argon-helium cryoablation
  Enhanced imaging examination (CT, MRI or color Doppler ultrasound)

SECONDARY OUTCOMES:
the iceball coverage rate during the procedure | during the procedure
  CT
Subjects' tolerance of the procedure | 1 week after the operation of argon-helium cryoablation
  questionnaire
the Eastern Cooperative Oncology Group Performance Status (ECOG PS) score | 4 weeks(±7d) after the operation of argon-helium cryoablation
  ECOG-PS questionnaire
To evaluate the operational performance of argon-helium cryoablation | during the procedure
  questionnaire